CLINICAL TRIAL: NCT04347889
Title: Prophylactic Hydroxychloroquine vs Vitamin C in Healthcare Workers at Risk of COVID-19: A RCT
Brief Title: Preventing COVID-19 in Healthcare Workers With HCQ: A RCT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Evidence that HCQ ineffective, loss of HCW interest,
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Professor and Vice Chairman for Research, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB2020-00222
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Covid-19
Keywords: covid-19; healthcare workers; prophylaxis; hydroxychloroquine
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Open label, controlled, RCT
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be masked to study assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (Experimental): Oral loading dose of 800 mg followed by once weekly oral hydroxychloroquine 400 mg for 3 months
  Interventions: Drug: Hydroxychloroquine
- Vitamin C (Active Comparator): Oral Vitamin C 1,000 mg daily for three months
  Interventions: Other: Vitamin C

INTERVENTIONS:
Drug: Hydroxychloroquine — Oral loading dose followed by once weekly dosing
  Arms: Hydroxychloroquine
Other: Vitamin C — Once daily vitamin C 1 gm
  Arms: Vitamin C

SUMMARY:
Healthcare workers (HCW) at risk of Covid-19 will have baseline serology for SARS-CoV-2 to see if they are already immune to Covid-19. HCW will get baseline assessment and if meeting inclusion criteria and no exclusion criteria they will be randomized in a 2:1 ratio to hydroxychloroquine or Vitamin C on a weekly basis for three months. Subjects will complete daily diary of symptoms and temperature, and will have repeat SARS-CoV-2 serology at 6 weeks and 3 months to determine seroconversion.

DETAILED DESCRIPTION:
Healthcare workers (HCW) at risk of Covid-19 will have baseline serology for SARS-CoV-2 to see if they are already immune to Covid-19. HCW will get baseline assessment and if meeting inclusion criteria and no exclusion criteria they will be randomized in a 2:1 ratio to hydroxychloroquine or Vitamin C on a weekly basis for three months. Subjects will complete daily diary of symptoms and temperature, and will have repeat SARS-CoV-2 serology at 6 weeks and 3 months to determine seroconversion.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker at risk of Covid-19

Exclusion Criteria:

* Known hypersensitivity or allergic reactions to 4-aminoquinoline compounds or its ingredients.
* Current, or history of, ocular macular disease or retinal damage.
* Current, or history of, subnormal glomerular filtration.
* Current use of tamoxifen citrate.
* Current, or history of, cardiomyopathy, atrial, nodal, or ventricular arrhythmias, torsades de pointes, conduction disorders (bundle branch block/atrio-ventricular heart block) or biventricular hypertrophy.
* Subjects taking other drugs that have the potential to prolong QT interval if taken with HCQ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Seroconversion rate | 3 months
  Percentage of healthcare worker who develop antibodies to SARS-CoV-2

SECONDARY OUTCOMES:
Admission for Covid-19 | 3 months
  Percentage of study subjects who require admission to a hospital for Covid-19